CLINICAL TRIAL: NCT03954717
Title: Pilot Study Evaluating Functional and Wellness Outcomes of the Shepherd CAN DO MS Program
Status: Completed | Type: Observational
Sponsor: Shepherd Center, Atlanta GA (Other)
Collaborators: Genzyme, a Sanofi Company (Industry); Can Do Multiple Sclerosis (Unknown)
Responsible Party: Principal Investigator, Deborah Backus, Director of Multiple Sclerosis Research, Shepherd Center, Atlanta GA
Other Study IDs: 1371420
Record Dates: First submitted 2019-05-14; First posted 2019-05-17 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Participants in the Shepherd CAN DO Program: People with MS enrolled into the Shepherd CAN DO Program.
  Interventions: Behavioral: Shepherd CAN DO Program
- Control Group-Shepherd (CG-S): People with MS who are current patients of the MS Institute at the Shepherd Center.
- Control Group-iConquerMS (CG-iCMS): iConquerMS members
- Support partners of CAN DO: Support partners of the participants in the Shepherd CAN DO Program group
  Interventions: Behavioral: Shepherd CAN DO Program
- CG-S support partners: Support partners of the people with MS in the CG-S group.
- CG-iCMS: Support partners of the people with MS in the CG-iCMS group

INTERVENTIONS:
Behavioral: Shepherd CAN DO Program — CAN DO Shepherd is a four-day participatory program held at the Shepherd Center, in Atlanta, Georgia or people with MS. The four-day program comprises evidence-based, comprehensive, and personalized educational and experiential opportunities aimed at empowering and enabling a person with MS to live a health life beyond their MS.
  Groups: Participants in the Shepherd CAN DO Program; Support partners of CAN DO

SUMMARY:
The study evaluates the efficacy of the CAN DO Program for improving health, wellness, and quality of life in people with MS, and compares outcomes between people with MS who participate in the CAN DO Program to a control group of people with MS who do not participate in the CAN DO Program. The study also evaluates the impact of the CAN DO Program on support partners.

DETAILED DESCRIPTION:
Can Do MS Programs offer evidence-based, comprehensive, and personalized educational and experiential opportunities aimed at empowering and enabling a person with MS to live a healthy life beyond their MS. The signature program of Can Do MS is the four-day CAN DO® Program (CAN DO). Preliminary outcomes suggest that participation in CAN DO leads to significant improvements in self-efficacy and various aspects of health status.1 The majority of 129 participants who participated in one of the three CAN DO Programs showed improvements in self-efficacy at one month (n=98), 3 months (n=84), and 6 months after the program (n=82; all p<0.001). Participants also showed significant improvements to varying degrees in subscales of the SF-36, including Physical Functioning (p=0.01), Role Physical, General Health, Vitality and Mental Health. These improvements were maintained to varying extents at one and 3 months post-program.

These important outcomes have not yet been compared to those in people with MS who receive traditional care but do not participate in this comprehensive educational opportunity. Furthermore, the impact on physical activity, participation, and quality of life has not been measured or compared to those who do not participate in CAN DO. Finally, recognizing the tremendous burden that can be placed on the support partner living and supporting a person with MS, education for support partners is another critical element of CAN DO. However, the impact on the support partner of empowering an individual with MS to adopt healthy behaviors also has not been assessed.

This project will allow Shepherd Center and Can Do MS to gather long-term health, wellness, and quality of life outcomes in people with MS and their support partners, as well as pilot data evaluating this study design for future larger scale clinical trials. Demonstrating the efficacy of this program will provide evidence that will impact the lives of people with MS and their families, specifically, their ability to live healthy lives independent of their MS.

ELIGIBILITY:
Inclusion Criteria:

* CAN DO Program group: have MS and participated in the May 2019 Shepherd CAN DO Program
* CG-iCMS: Have MS

Exclusion Criteria:

* CAN DO Program group: Active members of the Shepherd Center MS Wellness Program, or who have previously been a participant in any CAN DO MS Programs.
* CG-iCMS: Cannot participate in any of the CAN DO MS Programs at any time prior to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Twenty-four people with MS and their support partners participating in the May 2019 Shepherd CAN DO Program, and two control groups (CG) matched to program participants for age, sex, type of MS, and level of disability:
  CG-S = 24 current patients of the MS Institute at Shepherd and their support partners willing to complete surveys via an electronic platform.
  CG-iCMS = 24 iConquerMS members and their support partners willing to complete the same outcomes. These participants can be from anywhere in the US, but cannot participate in any of the Can Do MS programs at any time prior to the study.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Change in self-efficacy for symptom management at 6 months | 6 months
  The extent to which participants demonstrate increased self-efficacy (the confidence in one's belief to undertake a task) to manage symptoms measured by the Multiple Sclerosis Self-Management Scale Revised (MSSM-R)
  Constructs measured:
  * Healthcare provider relationship & communication
  * Treatment adherence/barriers
  * Social/family support
  * MS knowledge & information
  * Health maintenance behavior 24 items, with score 1 (disagree completely) to 5 (agree completely) For some 1 is a positive outcome and for others 5 is a positive outcome; the scores and transformed and scaled for each participant
Change in self-efficacy for symptom management at 12 months | 12 months
  The extent to which participants demonstrate increased self-efficacy (the confidence in one's belief to undertake a task) to manage symptoms measured by the Multiple Sclerosis Self-Management Scale Revised (MSSM-R)
  Constructs measured:
  * Healthcare provider relationship & communication
  * Treatment adherence/barriers
  * Social/family support
  * MS knowledge & information
  * Health maintenance behavior 24 items, with score 1 (disagree completely) to 5 (agree completely) For some 1 is a positive outcome and for others 5 is a positive outcome; the scores and transformed and scaled for each participant
Change in self-efficacy for symptom management at 24 months | 24 months
  The extent to which participants demonstrate increased self-efficacy (the confidence in one's belief to undertake a task) to manage symptoms measured by the Multiple Sclerosis Self-Management Scale Revised (MSSM-R)
  Constructs measured:
  * Healthcare provider relationship & communication
  * Treatment adherence/barriers
  * Social/family support
  * MS knowledge & information
  * Health maintenance behavior 24 items, with score 1 (disagree completely) to 5 (agree completely) For some 1 is a positive outcome and for others 5 is a positive outcome; the scores and transformed and scaled for each participant
Change in self-efficacy for quality of life at 6 months | 6 months
  The extent to which self-efficacy to undertake tasks related to quality of life increases over time as measured by the Exercise Self-Efficacy Scale (ESES) The Exercise Self-Efficacy Scale assesses an individual's beliefs in their ability to continue exercising on a three time per week basis at moderate intensities for 40+ minutes per session in the future. For each item, participants indicate their confidence to execute the behavior on a 100-point percentage scale comprised of 10-point increments, ranging from 0% (not at all confident) to 100% (highly confident). Total strength for each measure of self-efficacy is then calculated by summing the confidence ratings and dividing by the total number of items in the scale, resulting in a maximum possible efficacy score of 100.
Change in self-efficacy for quality of life at 12 months | 12 months
  The extent to which self-efficacy to undertake tasks related to quality of life increases over time as measured by the Exercise Self-Efficacy Scale (ESES) The Exercise Self-Efficacy Scale assesses an individual's beliefs in their ability to continue exercising on a three time per week basis at moderate intensities for 40+ minutes per session in the future. For each item, participants indicate their confidence to execute the behavior on a 100-point percentage scale comprised of 10-point increments, ranging from 0% (not at all confident) to 100% (highly confident). Total strength for each measure of self-efficacy is then calculated by summing the confidence ratings and dividing by the total number of items in the scale, resulting in a maximum possible efficacy score of 100.
Change in self-efficacy for quality of life at 24 months | 24 months
  The extent to which self-efficacy to undertake tasks related to quality of life increases over time as measured by the Exercise Self-Efficacy Scale (ESES) The Exercise Self-Efficacy Scale assesses an individual's beliefs in their ability to continue exercising on a three time per week basis at moderate intensities for 40+ minutes per session in the future. For each item, participants indicate their confidence to execute the behavior on a 100-point percentage scale comprised of 10-point increments, ranging from 0% (not at all confident) to 100% (highly confident). Total strength for each measure of self-efficacy is then calculated by summing the confidence ratings and dividing by the total number of items in the scale, resulting in a maximum possible efficacy score of 100.

SECONDARY OUTCOMES:
Change in caregiver perception of burden at 6 months | 6 months
  The extent to which caregivers of participants demonstrate decreased perception of caregiver burden as measured by the Zarit Burden Interview (ZBI) The ZBI consists of 22 items rated on a 5-point Likert scale that ranges from 0 (never) to 4 (nearly always) with the sum of scores ranging between 0-88. 9. Higher scores indicate greater burden. A score of 17 or more was considered high burden.
Change in caregiver perception of burden at 12 months | 12 months
  The extent to which caregivers of participants demonstrate decreased perception of caregiver burden as measured by the Zarit Burden Interview (ZBI) The ZBI consists of 22 items rated on a 5-point Likert scale that ranges from 0 (never) to 4 (nearly always) with the sum of scores ranging between 0-88. 9. Higher scores indicate greater burden. A score of 17 or more was considered high burden.
Change in caregiver perception of burden at 24 months | 24 months
  The extent to which caregivers of participants demonstrate decreased perception of caregiver burden as measured by the Zarit Burden Interview (ZBI) The ZBI consists of 22 items rated on a 5-point Likert scale that ranges from 0 (never) to 4 (nearly always) with the sum of scores ranging between 0-88. 9. Higher scores indicate greater burden. A score of 17 or more was considered high burden.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Backus, PhD, PT, Principal Investigator — Shepherd Center, Atlanta GA
Locations (1):
- Shepherd Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No